CLINICAL TRIAL: NCT06602505
Title: Comparative Analysis of Incidence of Newly Developed Postoperative Low Back Pain with Field Block Versus Without Field-block Before Spinal Anaesthesia for Patients Undergoing Caesarean Sections.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tata Main Hospital (Other)
Responsible Party: Principal Investigator, Dr.Deb Sanjay Nag, HOD & Head Consultant Anaesthesiology, Tata Main Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2222100059
Record Dates: First submitted 2024-09-15; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Caesarean Section
Keywords: Cesarean Section; Back Pain; Anesthesia, Local; Anesthesia, Spinal; Lidocaine
MeSH Terms: conditions — Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The person assessing the pain scores and the other observation parameters in the postoperative period was blinded to the group to which the patient was assigned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group B: No-field Block Group (No Intervention): Group B did not receive any field block before institution of subarachnoid block using 27 G Quincke's spinal needle for lower segment Caesarean section.
- Group A: Field Block Group (Experimental): Patients received field block with 5ml of 2% Lignocaine using a 24 G hypodermic needle before institution of subarachnoid block using 27 G Quincke's spinal needle for lower segment Caesarean section.
  Interventions: Procedure: Group A: Field Block Group

INTERVENTIONS:
Procedure: Group A: Field Block Group — Patients received field block with 5ml of 2% Lignocaine using a 24 G hypodermic needle before institution of subarachnoid block using 27 G Quincke's spinal needle for lower segment Caesarean section.
  Arms: Group A: Field Block Group

SUMMARY:
The study aimed to evaluate the effectiveness of field block in preventing postoperative low back pain (PDPB) in patients undergoing Cesarean Sections.

DETAILED DESCRIPTION:
The purpose of this study was to evaluate the effectiveness of field block with lidocaine 2% (5 ml) administered with a 24G hypodermic needle before spinal anesthesia for patients undergoing LSCS, in preventing the development of postoperative low back pain (PDPB). The study aimed to determine if using a field block would decrease the incidence of PDPB compared to patients who received only spinal anesthesia.

ELIGIBILITY:
Inclusion Criteria: All patients undergoing LSCS under spinal anesthesia, ASA Grade 2 and Grade 2E and willing to participate in the trial

Exclusion Criteria: Spine pathology/instability and coagulopathy, ASA Grade 3 and above, Pre-exiting low back pain, Morbid Obesity (BMI > 35), Patients needing more than 1 attempt for administration of spinal anaesthesia, Patients utilizing labour analgesia, Local infection or inflammation at the site of spinal anesthesia/field block, Unwilling to participate

-

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Only female patients, aged 18-45 years, posted for emergency or elective lower segment cesaerian section surgery
Enrollment: 220 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Incidence of postoperative back pain | 90 days
  Post operative back pain was assessed using a questionnaire specifically designed to evaluate back pain and transient neurological symptoms (e.g., unilateral or bilateral pain or radicular pain in the buttock, thigh, calves, or legs). Twenty-four hours after surgery, the patients were assessed for incidence and level of low back pain. In patients with back pain, the characteristics, aggravating factors, and degree of back pain was assessed using a numeric NRS. The same questionnaire was used telephonically to assess pain at 7 days, 1 month and 3 months after surgery.

SECONDARY OUTCOMES:
Birth weight of the child | 1 day
  Birth weight of the Child was measured at the birth of the baby
Period of gestation (weeks) | Weeks between conception and birth when a baby through Caesarean Section
  The period of gestation is the time between conception and birth when a baby through Caesarean Section in this study.
Gravida | 1 day
  Gravida at the time of Caesarean. It refers to a woman who is pregnant or has been pregnant in the past, regardless of the outcome of the pregnancy.

CONTACTS AND LOCATIONS:
Locations (1):
- Tata Main Hospital, Jamshedpur, Jharkhand, India

IPD SHARING:
Plan to Share IPD: Undecided
Being a GDPR compliant organization, permission of the Data Security Officer has to be obtained. However, masked data may be considered and provided if approved by the organization.